CLINICAL TRIAL: NCT03060525
Title: Deaf Weight Wise 2.0: Clinical Trial of a Healthy Lifestyle Intervention With Deaf Adults Ages 21 to 70
Brief Title: Deaf Weight Wise 2.0: A Healthy Lifestyle Intervention With Deaf Adults Who Are Overweight or Obese
Acronym: DWW2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Steve Barnett, Director, Rochester Prevention Research Center, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Deaf Weight Wise 2.0
Record Dates: First submitted 2017-02-18; First posted 2017-02-23 (Actual); Results first posted 2024-07-05 (Actual); Last update posted 2024-07-05 (Actual); Status verified 2024-01

CONDITIONS: Overweight; Obesity
Keywords: Deaf; American Sign Language; Overweight; Obese
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Immediate Group Intervention (Experimental): This arm will receive the DWW 2.0 Group intervention in Year 1 of the clinical trial. The group intervention will consist of groups of approximately 6-8 subjects who meet together for 16 weeks, for two hours each week. A trained, deaf, American Sign Language (ASL)-fluent DWW 2.0 counselor will lead the sessions. Subjects will be asked to complete a daily food and physical activity diary during the course of the 16-week intervention. Each intervention session will include a weigh-in, group sharing and problem solving, discussion of a weight management topic, which may include watching a powerpoint presentation and/or video; and a discussion on goal setting and action planning for the next week.
  Interventions: Behavioral: Deaf Weight Wise 2.0
- Immediate Videophone Intervention (Experimental): This arm will receive the DWW 2.0 Individual Videophone intervention in Year 1 of the clinical trial. The participant and their intervention counselor will have one-on-one sessions that take place via videophone (like a Skype call), for one hour each week. Each session will be led by a trained deaf, ASL-fluent DWW 2.0 counselor and will be held at a scheduled appointment time that is agreed upon by the subject and the counselor. Subjects will be asked to complete a daily food and physical activity diary during the course of the 16-week intervention. Each intervention session will include a weigh-in, personal sharing and problem solving, discussion of a weight management topic, which may include watching a powerpoint presentation and/or video; and a discussion on goal setting and action planning for the next week.
  Interventions: Behavioral: Deaf Weight Wise 2.0
- Delayed Group Intervention (Other): This arm will receive the DWW 2.0 Group intervention in Year 2 of the clinical trial. The group intervention will consist of groups of approximately 6-8 subjects who meet together for 16 weeks, for two hours each week. A trained, deaf, American Sign Language (ASL)-fluent DWW 2.0 counselor will lead the sessions. Subjects will be asked to complete a daily food and physical activity diary during the course of the 16-week intervention. Each intervention session will include a weigh-in, group sharing and problem solving, discussion of a weight management topic, which may include watching a powerpoint presentation and/or video; and a discussion on goal setting and action planning for the next week.
  Interventions: Behavioral: Deaf Weight Wise 2.0
- Delayed Videophone Intervention (Other): This arm will receive the DWW 2.0 Individual Videophone intervention in Year 2 of the clinical trial. The participant and their intervention counselor will have one-on-one sessions that take place via videophone (like a Skype call), for one hour each week. Each session will be led by a trained deaf, ASL-fluent DWW 2.0 counselor and will be held at a scheduled appointment time that is agreed upon by the subject and the counselor. Subjects will be asked to complete a daily food and physical activity diary during the the course of the 16-week intervention. Each intervention session will include a weigh-in, personal sharing and problem solving, discussion of a weight management topic, which may include watching a powerpoint presentation and/or video; and a discussion on goal setting and action planning for the next week.
  Interventions: Behavioral: Deaf Weight Wise 2.0

INTERVENTIONS:
Behavioral: Deaf Weight Wise 2.0 — Deaf Weight Wise 2.0 is a group or individual intervention lead by trained, American Sign Language fluent Deaf counselors, who utilize an existing evidence-based curriculum that emphasizes healthy eating, exercise, and lifestyle components. It is a behavior change intervention that uses motivational interviewing techniques to help participants identify/recognize their own unhealthy behaviors, help individuals build skills that will promote behavior change, and help group members to support each other to make behavior changes. The Curriculum includes group exercise activities ("Do It!"), experiential learning activities ("Try It!" such as learning how to read a nutrition label or modify a recipe to make it healthier), and group activities related to food preparation or sampling healthy foods ("Taste It!"). Self-monitoring using daily food diaries and weekly "weigh-ins" is also a key component. The intervention also includes a 6-month follow up and maintenance phase.

SUMMARY:
The purpose of the Deaf Weight Wise 2.0 (DWW 2.0) study is to test an evidence-based, comprehensive program to modify obesity-related health behaviors with Deaf people ages 21 to 70 who use American Sign Language (ASL) as their primary language. Participants will be randomized to one of four arms: immediate intervention vs. intervention delayed one year, and in-person group intervention vs. individual intervention delivered via videophone. The investigators' primary hypothesis is that participants in the immediate DWW 2.0 intervention will increase their physical activity and reduce their caloric intake and body weight compared with those in the delayed intervention group (no intervention yet).

ELIGIBILITY:
Inclusion Criteria:

* Deaf men and women ages 21-70 years who use sign language and live in the Rochester Metropolitan Statistical Area (MSA),
* have a body mass index (BMI) of 25-45.
* Eligible subjects must also have permission to participate from a primary healthcare provider if: 1) self-reported diagnosis of a recent cardiovascular disease event (heart attack or stroke in past 6 months), 2) self-reported heart condition, chest pain, dizziness, or other reason not to participate in physical activity, 3) had weight loss surgery in the previous 2 years (self-reported), and 4) are pregnant (self-reported).
* Subjects must also be willing to follow a healthy dietary pattern and to abstain from using weight loss medications during the study, and be willing and able to attend either group or videophone sessions, and to participate in data collection requirements.

Exclusion Criteria:

* Exclusion criteria include: subjects without medical clearance who had 1) a cardiovascular disease event in the past six months, 2) or heart condition, chest pain, dizziness, or other reason not to participate in physical activity, 3) or weight loss surgery in the past two years, or 4) are pregnant. Participants with these conditions (as determined by the PAR-Q Physical Activity Readiness-Questionnaire and other questions administered during the initial study screening visit) must obtain medical clearance from their primary healthcare clinician (or maternity care clinician for pregnancy) to be eligible. Those who are unable or unwilling to provide written, informed consent, and inability to see and interact with computer-based questionnaires and educational interventions will be excluded.

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2017-01-25 (Actual); Primary Completion 2019-08-29 (Actual); Study Completion 2019-08-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven L Barnett, MD, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester; National Center for Deaf Health Research, Rochester, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study recruited participants using a variety of methods, and had a rolling enrollment (in 4 waves). The first participant was enrolled on Jan. 25, 2017 and the last participant was enrolled on Sept. 22, 2017.
Groups:
- Immediate Group Intervention: Participants received the DWW 2.0 Group intervention in Year 1 of the clinical trial. The group intervention consisted of groups of approximately 6-8 subjects who meet together for 16 weeks, for two hours each week. A trained, deaf, American Sign Language (ASL)-fluent DWW 2.0 counselor led the sessions. Subjects were asked to complete a daily food and physical activity diary during the course of the 16-week intervention. Each intervention session included a weigh-in, group sharing and problem solving, discussion of a weight management topic, and a discussion on goal setting and action planning for the next week.
  Deaf Weight Wise 2.0 is a group or individual intervention lead by trained, American Sign Language fluent Deaf counselors, who utilize an existing evidence-based curriculum that emphasizes healthy eating, exercise, and lifestyle components. It is a behavior change intervention that uses motivational interviewing techniques to help participants identify/recognize unhealthy behaviors, build skills that will promote behavior change, and help group members to support each other to make behavior changes. The Curriculum includes group exercise ("Do It!"), experiential learning ("Try It!" such as learning how to read a nutrition label), and group activities such as sampling healthy foods ("Taste It!"). Self-monitoring using daily food diaries and weekly "weigh-ins" are encouraged. The intervention also includes a 6-month follow up and maintenance phase.
- Immediate Videophone Intervention: Participants received the DWW 2.0 Individual Videophone intervention in Year 1 of the clinical trial. The participant and their intervention counselor had one-on-one sessions via videophone, for one hour each week. Each session was led by a trained deaf, ASL-fluent DWW 2.0 counselor. Subjects were asked to complete a daily food and physical activity diary during the course of the 16-week intervention. Each intervention session included a weigh-in, personal sharing and problem solving, discussion of a weight management topic, and a discussion on goal setting and action planning for the next week.
  Deaf Weight Wise 2.0 is a group or individual intervention lead by trained, American Sign Language fluent Deaf counselors, who utilize an existing evidence-based curriculum that emphasizes healthy eating, exercise, and lifestyle components. It is a behavior change intervention that uses motivational interviewing techniques to help participants identify/recognize unhealthy behaviors, build skills that will promote behavior change, and help group members to support each other to make behavior changes. The Curriculum includes group exercise ("Do It!"), experiential learning ("Try It!" such as learning how to read a nutrition label), and group activities such as sampling healthy foods ("Taste It!"). Self-monitoring using daily food diaries and weekly "weigh-ins" are encouraged. The intervention also includes a 6-month follow up and maintenance phase.
- Delayed Group Intervention: Participants received the DWW 2.0 Group intervention in Year 2 of the clinical trial. The group intervention consisted of groups of approximately 6-8 subjects who meet together for 16 weeks, for two hours each week. A trained, deaf, American Sign Language (ASL)-fluent DWW 2.0 counselor led the sessions. Subjects were asked to complete a daily food and physical activity diary during the course of the 16-week intervention. Each intervention session included a weigh-in, group sharing and problem solving, discussion of a weight management topic, and a discussion on goal setting and action planning for the next week.
  Deaf Weight Wise 2.0 is a group or individual intervention lead by trained, American Sign Language fluent Deaf counselors, who utilize an existing evidence-based curriculum that emphasizes healthy eating, exercise, and lifestyle components. It is a behavior change intervention that uses motivational interviewing techniques to help participants identify/recognize unhealthy behaviors, build skills that will promote behavior change, and help group members to support each other to make behavior changes. The Curriculum includes group exercise ("Do It!"), experiential learning ("Try It!" such as learning how to read a nutrition label), and group activities such as sampling healthy foods ("Taste It!"). Self-monitoring using daily food diaries and weekly "weigh-ins" are encouraged. The intervention also includes a 6-month follow up and maintenance phase.
- Delayed Videophone Intervention: Participants received the DWW 2.0 Individual Videophone intervention in Year 2 of the clinical trial. The participant and their intervention counselor had one-on-one sessions via videophone, for one hour each week. Each session was led by a trained deaf, ASL-fluent DWW 2.0 counselor. Subjects were asked to complete a daily food and physical activity diary during the course of the 16-week intervention. Each intervention session included a weigh-in, personal sharing and problem solving, discussion of a weight management topic, and a discussion on goal setting and action planning for the next week.
  Deaf Weight Wise 2.0 is a group or individual intervention lead by trained, American Sign Language fluent Deaf counselors, who utilize an existing evidence-based curriculum that emphasizes healthy eating, exercise, and lifestyle components. It is a behavior change intervention that uses motivational interviewing techniques to help participants identify/recognize unhealthy behaviors, build skills that will promote behavior change, and help group members to support each other to make behavior changes. The Curriculum includes group exercise ("Do It!"), experiential learning ("Try It!" such as learning how to read a nutrition label), and group activities such as sampling healthy foods ("Taste It!"). Self-monitoring using daily food diaries and weekly "weigh-ins" are encouraged. The intervention also includes a 6-month follow up and maintenance phase.
Period: Overall Study
Arm/Group | Immediate Group Intervention | Immediate Videophone Intervention | Delayed Group Intervention | Delayed Videophone Intervention
Started | 16 | 18 | 21 | 21
Completed | 13 | 14 | 17 | 18
Not Completed | 3 | 4 | 4 | 3
Not completed — moved out of state | 1 | 1 | 1 | 1
Not completed — unable to meet time commitment required of study | 2 | 3 | 3 | 1
Not completed — no longer interested in doing intervention | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Immediate Group Intervention | Immediate Videophone Intervention | Delayed Group Intervention | Delayed Videophone Intervention | Total
Number analyzed (Participants) | 16 | 18 | 21 | 21 | 76
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.3 (13.1) | 43.4 (13.4) | 38.9 (16.8) | 45.2 (15.4) | 42.4 (14.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 13 | 18 | 13 | 56
  Male | 4 | 5 | 3 | 8 | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 1 | 0 | 3
  Not Hispanic or Latino | 16 | 16 | 20 | 21 | 73
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 1 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 3 | 2 | 3 | 9
  White | 13 | 13 | 17 | 17 | 60
  More than one race | 0 | 1 | 1 | 0 | 2
  Unknown or Not Reported | 2 | 0 | 0 | 0 | 2
Age became deaf [Count of Participants; unit: Participants] — Self-reported age at which participant became deaf
  Participants
    Became deaf at age 3 or younger (including born deaf) | 14 | 17 | 18 | 20 | 69
    Became deaf at age 4 or older | 1 | 1 | 3 | 0 | 5
    Unknown | 1 | 0 | 0 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Change in Body Weight (kg)
Description: measure mean change = 6-month weight - baseline weight, for the immediate and delayed intervention groups (change from pre to post intervention).
Time Frame: 6 month weight (kg) - baseline weight (kg)
Population: 62 cases were included in analysis of primary outcomes (out of 76 enrolled). 14 cases were excluded from analysis because they had data for only one timepoint out of five timepoints.
Measure: Least Squares Mean (Standard Error); unit: kg
Arm/Group | Immediate Group Intervention | Immediate Videophone Intervention | Delayed Group Intervention | Delayed Videophone Intervention
Number analyzed (Participants) | 14 | 14 | 17 | 17
kg | -2.36 (1.56) | -3.09 (1.54) | 1.02 (1.49) | 0.26 (1.37)
Statistical Analysis 1: Comparison: Immediate Group Intervention vs Immediate Videophone Intervention vs Delayed Group Intervention vs Delayed Videophone Intervention; Difference in weight change from Baseline to 6months, between Immediate Intervention participants (group and videophone combined) vs. Delayed Intervention participants (group and videophone combined). [analysis of 2 arms, immediate intervention vs. delayed intervention]; Test type: Superiority; p = 0.026, Mixed Models Analysis; Mean Difference (Final Values) = -3.36, 95% CI 2-sided [-6.32 to -0.41], Standard Error of Mean 1.51

2. Primary Outcome: Change in BMI (Body Mass Index)
Description: measure mean change = 6-month BMI - baseline BMI, for the immediate and delayed intervention groups (change from pre to post intervention).
Time Frame: 6-month BMI - baseline BMI
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: kg/m^2
Arm/Group | Immediate Group Intervention | Immediate Videophone Intervention | Delayed Group Intervention | Delayed Videophone Intervention
Number analyzed (Participants) | 14 | 14 | 17 | 17
kg/m^2 | -0.91 (0.61) | -1.05 (0.60) | 0.39 (0.58) | 0.20 (0.53)
Statistical Analysis 1: Comparison: Immediate Group Intervention vs Immediate Videophone Intervention vs Delayed Group Intervention vs Delayed Videophone Intervention; Difference in Body Mass Index (BMI) change from Baseline to 6months, between Immediate Intervention participants (group and videophone combined) vs. Delayed Intervention participants (group and videophone combined). [analysis of 2 arms, immediate intervention vs. delayed intervention]; Test type: Superiority; p = 0.03, Mixed Models Analysis; Mean Difference (Final Values) = -1.27, 95% CI 2-sided [-2.42 to -0.12], Standard Error of Mean 0.59

3. Primary Outcome: Change in Physical Activity
Description: change in amount of physical activity = 6-month MET-minutes/week - baseline MET-minutes/week (change from pre to post intervention), using the International Physical Activity Questionnaire. IPAQ score is a continuous measure and reports median MET-minutes per week (a combination of walking met-minutes/week + moderate activity MET-minutes/week + vigorous activity MET-minutes/week).
Time Frame: 6-month MET-min/wk - baseline MET-min/wk
Population: 56 cases were included in analysis of this physical activity primary outcomes (out of 76 enrolled). 14 cases were excluded from analysis because they had data for only one timepoint out of five timepoints (76-14=62); an additional 6 cases were excluded from the physical activity analysis due to missing physical activity data at the 6-month time point (n=56 for analysis).
Measure: Median (Inter-Quartile Range); unit: MET-minutes/wk
Arm/Group | Immediate Group Intervention | Immediate Videophone Intervention | Delayed Group Intervention | Delayed Videophone Intervention
Number analyzed (Participants) | 12 | 13 | 14 | 17
MET-minutes/wk | 2.75 [-1658.00 to 839.25] | 543.50 [-174.00 to 786.00] | -82.50 [-1074.00 to 480.00] | 66.00 [-381.00 to 612.00]
Statistical Analysis 1: Comparison: Immediate Group Intervention vs Immediate Videophone Intervention vs Delayed Group Intervention vs Delayed Videophone Intervention; change in amount of physical activity = 6-month MET-minutes/week - baseline MET-minutes/week (change from pre to post intervention), using the International Physical Activity Questionnaire. IPAQ score is a continuous measure and reports median MET-minutes per week (a combination of walking met-minutes/week + moderate activity MET-minutes/week + vigorous activity MET-minutes/week). [analysis of 2 arms, immediate intervention vs. delayed intervention]; Test type: Superiority; p = 0.63, Wilcoxon (Mann-Whitney); Median Difference (Net) = 247.50

ADVERSE EVENTS:
Time Frame: Baseline (data point 1) to 24-month data collection point (final data point 5); total of 2 years.
Arm/Group | Immediate Group Intervention | Immediate Videophone Intervention | Delayed Group Intervention | Delayed Videophone Intervention
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/18 | 0/21 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/18 | 0/21 | 0/21
Other Adverse Events (participants affected / at risk) | 0/16 | 0/18 | 0/21 | 0/21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-10-17): https://cdn.clinicaltrials.gov/large-docs/25/NCT03060525/Prot_SAP_000.pdf